CLINICAL TRIAL: NCT02606123
Title: A Phase 1/2 Open-Label Study to Assess the Safety, Pharmacokinetics, and Anti-Tumor Activity of Oral EPI-506 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Safety and Anti-Tumor Study of Oral EPI-506 for Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At end of Phase 1 excessive high pill burden (18 capsules/day)
Sponsor: ESSA Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI-506-CS-0001
Record Dates: First submitted 2015-10-22; First posted 2015-11-17 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms, Male; Genital Diseases, Male; Prostatic Diseases
Keywords: Prostate Cancer; Metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Genital Diseases, Male; Prostatic Diseases | interventions — EPI-506

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-506 (Experimental): Part I: Ascending doses of EPI-506 administered orally to define the maximum tolerated dose.
  Interventions: Drug: EPI-506

INTERVENTIONS:
Drug: EPI-506 — Patients will receive EPI-506 as an oral softgel capsule.
  Part 1:
  Approximately six dose levels of EPI-506 will be studied, beginning at 80 mg/day. During the Single-Dose Period, patients will first receive a dose of EPI-506 in the fasted state followed by 2 days of washout, and then patients will receive a second dose of EPI-506 in the fed state followed by 2 days of washout. Patients will then enter the Multiple Dosing and Long-term Dosing Period where they will receive once or twice daily dosing in a fed or fasted state until they meet discontinuation criteria.
  Part 2:
  The dose in Part 2 will be determined in Part 1 of the study. Patients will receive the Part 2 dose daily until they meet discontinuation criteria.

SUMMARY:
The study will consist of 2 parts: Part I (Dose Escalation) and Part II (Dose Expansion). In Part I, patients will participate in single, multiple, and long-term dosing periods using EPI-506 to determine safety, pharmacokinetics, the maximum tolerated dose, and preliminary indications of anti-tumor activity. Part I is an open-label, adaptive 3 + 3 design, dose-escalation study. Approximately six dose levels of EPI-506 will be studied, beginning at 80 mg/day. Enrolled patients may be allowed to escalate to a subsequent dose cohort after their initial twelve weeks. Additional patients may be enrolled at any safe dose level prior to or concurrent with enrolling patients in Part II.

In Part II, 3 patient populations; post-abiraterone metastatic castration-resistant prostate cancer (mCRPC) but enzalutamide-naïve, post-enzalutamide mCRPC but abiraterone-naïve, and post-abiraterone and enzalutamide mCRPC will be studied at the recommended Phase 2 dose (RP2D) determined in Part I over 12 weeks of daily dosing. Approximately 120 patients (40 in each cohort) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the Prostate
* Metastatic Disease with at least one lesion on bone scan and/or soft tissue on CT/MRI
* Demonstrated progression on abiraterone and/or enzalutamide
* Demonstrated PSA progression within 12 weeks of study participation
* Castrate testosterone levels at screening with continued Luteinizing hormone-releasing hormone (LHRH) therapy
* Eastern Cooperative Oncology Group (ECOG) score between 0-1
* Asymptomatic or mildly symptomatic

Exclusion Criteria:

* Candidates for cytotoxic chemotherapy
* Received more than one line of chemotherapy
* Received more than one treatment course of enzalutamide or abiraterone
* Inadequate washout of prohibited hormonally active agents or other prior treatments for prostate cancer (PCa)
* Known intra-cerebral disease or brain mets
* Spinal cord compression within 6 months
* Prior treatment with investigative androgen receptor (AR) agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Part I: Safety and tolerability assessed by vital signs, laboratory measurements, and frequency and severity of treatment-related adverse events | 12 weeks
Part II: Prostate-specific antigen (PSA) response rate | 12 weeks

SECONDARY OUTCOMES:
Part I: Define the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) | 9 months
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by plasma area under the plasma concentration-time curve (AUC)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by maximum concentration (Cmax)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by observed pre-dose plasma concentration during multiple dosing (Ctrough)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by time to reach Cmax (tmax)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by apparent terminal elimination half-life (t1/2)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by apparent volume of distribution during the terminal phase after extravascular administration (Vz/F)
Part I: Pharmacokinetics (PK) profile of EPI-506 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by apparent clearance after extravascular administration (CL/F)
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by AUC
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by Cmax
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by Ctrough
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by tmax
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by t1/2
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by Vz/F
Part I: Pharmacokinetics (PK) profile of EPI-002 | Pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, 24h, and 48h after dose; Day 8 at pre-dose, and at 15min, 30min 1h, 2h, 4h, 6h, 8h, 12h, 24h after dose.
  Assessed by CL/F
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by AUC
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by Cmax
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by Ctrough
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by tmax
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by t1/2
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by Vz/F
Part I: Food effect on PK | 6 days
  Following a single-dose of EPI-506 on Days 1 and 4 assessed by CL/F
Part I: PSA | Baseline to Week 12
  Evaluated as a Pharmacodynamic (PD) marker of response
Part II: Safety and tolerability assessed by vital signs, laboratory measurements, and frequency and severity of treatment-related adverse events | 12 months
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by AUC
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Cmax
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Ctrough
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by tmax
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by t1/2
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Vz/F
Part II: To evaluate the PK of EPI-506 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by CL/F
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by AUC
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Cmax
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Ctrough
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by tmax
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by t1/2
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by Vz/F
Part II: To evaluate the PK of EPI-002 | Day 8 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, 8h, 12h, and 24h after dose; Week 12 at pre-dose, and at 15min, 30min, 1h, 2h, 4h, 6h, and 8h after dose.
  Assessed by CL/F
Part II: Time to PSA progression | 12 months
Part II: Radiographic progression | 12 weeks
  Radiographic progression evaluated per modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1
Part II: Objective response | 12 weeks
  Radiographic progression evaluation per mRECIST v1.1 in patients with measurable soft tissue disease at baseline

OTHER OUTCOMES:
Exploratory Objective: Biomarkers | 12-24 months
  Circulating tumor cells (CTCs) with emphasis on androgen receptor splice variants (AR-V7)
Exploratory Objective: Pain assessments | 12-24 months
  Assessed by Brief Pain Inventory-Short Form (BPI-SF) instrument

CONTACTS AND LOCATIONS:
Overall Officials: Frank Perabo, MD, PhD, Study Director — ESSA Pharmaceuticals Corp.; Robert B. Montgomery, MD, Principal Investigator — Seattle Cancer Care Alliance; Kim N. Chi, MD, Principal Investigator — British Columbia Cancer Agency - Vancouver Centre
Locations (5):
- United States (4):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Seattle Cancer Care Alliance, Seattle, Washington
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada